CLINICAL TRIAL: NCT06693908
Title: A Phase Ic Open-label Study to Evaluate the Pharmacodynamic Effects, Pharmacokinetics, and Safety of Vixarelimab in Patients With Moderate to Severe Active Ulcerative Colitis
Brief Title: A Study to Evaluate the Activity, and Safety of Vixarelimab in Participants With Moderate to Severe Active Ulcerative Colitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA45735; 2024-516287-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Ulcerative Colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vixarelimab (Experimental): Participants will receive subcutaneous (SC) injections of vixarelimab during the treatment period.
  Interventions: Drug: Vixarelimab

INTERVENTIONS:
Drug: Vixarelimab — Vixarelimab will be administered as per the schedule specified.
  Other Names: RO7622888; KPL-716

SUMMARY:
This study aims to evaluate the pharmacodynamic (PD) effects of vixarelimab in the gut of participants with active moderate to severe ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC established at least 3 months
* Moderately to severely active UC
* Participants must meet criteria for either advanced therapy failure or conventional therapy failure

Exclusion Criteria:

* Diagnosis of Crohn's disease or indeterminate colitis
* Suspicion of ischemic colitis, radiation colitis, microscopic colitis or infectious colitis
* Prior colectomy
* Prior treatment with systemic janus kinase (JAK) inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Fibroblast Products From Colonic Tissue | Baseline up to approximately 3 months

SECONDARY OUTCOMES:
Serum Concentration of Vixarelimab | Up to approximately 3 months
Number of Participants with Anti-drug Antibodies (ADA) to Vixarelimab | Up to approximately 3 months
Number of Participants With Adverse Events (AEs), With Severity Determined According to Division of AIDS (DAIDS) Toxicity Grading Scale | Up to approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No